CLINICAL TRIAL: NCT05941520
Title: Phase IIA Trial of Acolbifene (20 mg) vs Low Dose Tamoxifen (5 mg) in Pre-menopausal Women at High Risk for Development of Breast Cancer
Brief Title: Acolbifene Versus Low Dose Tamoxifen for the Prevention of Breast Cancer in Premenopausal Women at High Risk for Development of Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2023-05217; NCI-2023-05217 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UMCC 2022.055 (Other: University of Michigan Rogel Cancer Center); UMI22-09-01 (Other: DCP); P30CA046592 (NIH); UG1CA242632 (NIH)
Record Dates: First submitted 2023-07-11; First posted 2023-07-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Breast Atypical Hyperplasia; Breast Carcinoma; Breast Ductal Carcinoma In Situ; Breast Lobular Carcinoma In Situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Specimen Handling; Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (acolbifene) (Experimental): Patients receive acolbifene PO QD for 6 months in the absence of disease progression or unacceptable toxicity. Patients also undergo 3D mammography and collection of blood samples during screening and at the end of acolbifene treatment. In addition, patients undergo RPFNA during screening and during day 1-10 of their menstrual cycle, or if not menstruating, at the convenience of the patient and study staff.
  Interventions: Drug: Acolbifene Hydrochloride; Procedure: Biospecimen Collection; Other: Questionnaire Administration; Procedure: Random Periareolar Fine-Needle Aspiration
- Group 2 (tamoxifen) (Active Comparator): Patients receive tamoxifen PO QD for 6 months in the absence of disease progression or unacceptable toxicity. Patients also undergo 3D mammography and collection of blood samples during screening and at the end of tamoxifen treatment. In addition, patients undergo RPFNA during screening and day 1-10 of their menstrual cycle, or if not menstruating, at the convenience of the patient and study staff.
  Interventions: Procedure: Biospecimen Collection; Procedure: Mammography; Other: Questionnaire Administration; Procedure: Random Periareolar Fine-Needle Aspiration; Drug: Tamoxifen

INTERVENTIONS:
Drug: Acolbifene Hydrochloride — Given PO
  Arms: Group 1 (acolbifene)
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Mammography — Undergo 3D mammography
  Other Names: MG
  Arms: Group 2 (tamoxifen)
Other: Questionnaire Administration — Ancillary studies
Procedure: Random Periareolar Fine-Needle Aspiration — Undergo RPFNA
  Other Names: Random Periareolar Fine Needle Aspiration; RPFNA
Drug: Tamoxifen — Given PO
  Other Names: TMX
  Arms: Group 2 (tamoxifen)

SUMMARY:
This phase IIA trial compares the effect of acolbifene versus low dose tamoxifen in preventing breast cancer in premenopausal women at high risk for developing breast cancer. The usual approach for patients at increased risk for breast cancer is to undergo yearly breast magnetic resonance imaging or ultrasound in addition to yearly mammogram. Premenopausal women at very high lifetime risk for breast cancer (greater than 50%) can consider preventive removal (mastectomy) of both breasts. Premenopausal women age 35 or older with a prior diagnosis of atypical hyperplasia, lobular carcinoma in situ, or an estimated 10-year risk of greater than or equal to 3% or estimated 10-year risk of greater than or equal to 2-5 times that of the average woman (depending on age) may be advised to consider five years of standard dose tamoxifen. Standard dose tamoxifen is four times the dose used in this study. Estrogen can cause the development and growth of breast cancer cells. Acolbifene and tamoxifen blocks the use of estrogen by breast cells. This study may help researchers measure the effects of acolbifene and low dose tamoxifen on markers of breast cancer risk in mammogram imaging, breast tissue, and in blood samples.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if there is a difference in change in expression of the endocrine resistance gene anterior gradient 2 (AGR2) in benign breast tissue of premenopausal women at increased risk for breast cancer randomized to acolbifene 20 mg versus (vs) tamoxifen 5 mg orally daily for 6 months.

SECONDARY OBJECTIVES:

I. To determine if there is significant within-arm effect of 6 months of acolbifene 20 mg or tamoxifen 5 mg as assessed on the Estrogen Response Gene Index (ERGI) in benign breast tissue.

II. To determine if there is significant within-arm effect of 6 months of acolbifene 20 mg or tamoxifen 5 mg on mammographic density as measured by change in fibroglandular volume (FGV) and mammographic percent dense volume.

III. To determine if there is a significant within-arm effect of 6 months of acolbifene 20 mg or tamoxifen 5 mg on Menopause-Specific Quality of Life Questionnaire (MENQOL) or Hot Flash Score.

EXPLORATORY OBJECTIVES:

I. Assess within arm change in breast epithelial cell protein expression of Ki-67 in specimens with >= 2% baseline Ki-67.

II. Assess within arm change in bioavailable serum estradiol, testosterone, progesterone.

III. Association of baseline anti-Mullerian hormone (AMH) (>= 1 ng/ml associated with normal ovarian reserve) with 6-month serum estradiol and change in tissue estrogen responsive gene expression (ERGI and AGR2).

IV. Association of tamoxifen and acolbifene parent drug and active metabolite levels with change in tissue estrogen response genes and mammographic density.

V. Assess within arm change of AGR2, Forkhead box protein A1 (FOXA1), estrogen receptor (ER), progesterone receptor (PR) proteins on residual fixed specimens acquired by random periareolar fine needle aspiration (RPFNA) and processed to blocks.

VI. Assess within arm change in metabolic measures including triglycerides, measures of insulin sensitivity and thyroid binding globulin (Kansas University Medical Center [KUMC] participants only).

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive acolbifene orally (PO) once daily (QD) for 6 months in the absence of disease progression or unacceptable toxicity. Patients also undergo three-dimensional (3D) mammography and collection of blood samples during screening and at the end of acolbifene treatment. In addition, patients undergo RPFNA during screening and on day 1-10 of their menstrual cycle, or if not menstruating, at the convenience of the patient and study staff.

GROUP II: Patients receive tamoxifen PO QD for 6 months in the absence of disease progression or unacceptable toxicity. Patients also undergo 3D mammography and collection of blood samples during screening and at the end of tamoxifen treatment. In addition, patients undergo RPFNA during screening and day 1-10 of their menstrual cycle, or if not menstruating, at the convenience of the patient and study staff.

After completion of study treatment, patients are followed up between 21-35 days.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 35 years
* Considered clinically premenopausal
* Having regular menstrual cycles (between 21 and 35 days) unless a contraceptive device such as progestin containing intrauterine device (IUD) (e.g., Mirena IUD) is being used which suppresses menstrual periods, or premenopausal women who have undergone a hysterectomy, but ovaries are intact
* Not considering pregnancy for at least 12 months
* Women of child-bearing potential capacity must be willing to have used effective birth control precautions for 8 weeks prior to fine needle aspiration and be willing to continue for 8 weeks after study completion as tamoxifen may have teratogenic effects on the developing fetus. Reproductive and developmental toxicity studies have not been conducted with acolbifene. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must stop study drug and inform her study physician immediately.

  * For women not using oral contraceptive (progestin alone or estrogen plus a progestin), two of the following are recommended but woman must agree to at least one of the following methods:

    * IUD non-hormonal or hormone containing (usually a progestin) intrauterine device (IUD) or rings. Any of these should have been inserted at least 8 weeks prior to RPFNA.
    * Barrier method (such as condoms and diaphragms or cervical caps with or without a spermicide)
    * Partner has had a vasectomy.
  * For women using oral contraceptive (progestin alone or estrogen plus a progestin), woman must agree to at least a non- hormonal IUD or a barrier method (below) or her partner must have had a vasectomy:

    * Non-hormonal IUD
    * Barrier method (such as condoms and diaphragms or cervical caps with or without a spermicide)
    * Partner has had a vasectomy
* Must have increased breast cancer risk as predicted by any one or more of the conditions listed below or increased model calculated risk as below:

  * Any one or more of the following conditions associated with increased risk (condition must be documented in electronic medical record or copy of relevant pathology or genetic testing reports submitted with the eligibility checklist)

    * A prior biopsy at any time in the past showing ductal carcinoma in situ (DCIS), lobular carcinoma in situ (LCIS), atypical hyperplasia. (If DCIS must have been treated by mastectomy or local excision +/- radiation with this treatment completed at least 3 months prior to screening with RPFNA)
    * High or moderate penetrance risk pathogenic or likely pathogenic germline gene mutation in ATM, BARD1, BRIP1, CDH1, CHEK2, MSH6, NBN, NF1, PTEN, PMS2, RAD51C, RAD51D, or TP53
    * High polygenic risk score (Life-time risk of >= 2x average or 25%)
    * Breast cancer in a first or second degree relative (female or male) with onset under age 50. First degree relative is defined as parent, sibling, or child. Second degree relative is defined as grandparent, uncle, aunt, nephew, niece, half-sibling, grandchild or first cousin
    * Two or more affected first or second-degree relatives from either the maternal or paternal lineage without regard to age
    * Bilateral breast cancer or breast and ovarian cancer in the same first or second degree relative without regard to age.
    * High mammographic density defined as either visual estimate of area of density (VAS) > 50%, or Volpara (Trademark) >= 15% dense volume (Volpara d) or Breast Imaging Reporting and Data System (BIRADS) assessment of extremely dense (BIRADs D)
  * Alternatively, instead of conditions listed above, an increased risk of breast cancer as calculated by International Breast Cancer Intervention Study Version 8 (IBIS 8), or Breast Cancer Surveillance Consortium (BCSC) 3 by one or more of the following criteria:

    * 10-year risk of breast cancer of >= 3%
    * Increase in age specific 10-year relative risk by age group

      * Age 35-39 10-year relative risk of >= 5X that for age group
      * Age 40-44 10-year risk of >= 4X that for age group
      * Age 45 and up 10-year risk of >= 2X
    * IBIS Version 8 Remaining lifetime risk of >= 25% or >= 2X that of population
  * A copy of the output of model calculations from IBIS 8 (https://ems-trials.org/riskevaluator/), or BCSC version 3.0 (https://tools.bcsc-scc.org/BC5yearRisk/calculator.htm) online tools, if used for qualifying risk assessment, or polygenetic risk score should be submitted with the eligibility checklist. Otherwise, these risk qualifying factors need to be documented in the medical record if that is considered the source document
* Women must have at least 1 unaffected untreated breast for fine needle aspiration. Women may have had prior unilateral breast radiation or mastectomy for DCIS
* Eastern Cooperative Oncology Group (ECOG) current performance status (PS) ≤ 2 as documented within 3 months prior to randomization or Karnofsky score >= 60%
* Total bilirubin =< 1.5 x institutional upper limit of normal (measured within 180 days prior to randomization)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 1.5 x institutional upper limit of normal (measured within 180 days prior to randomization)
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 x institutional upper limit of normal (measured within 180 days prior to randomization)
* Creatinine =< 2.0 mg/dL (measured within 180 days prior to randomization)
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Bilateral breast implants (danger of implant puncture with RPFNA)
* Women who are pregnant
* Currently breastfeeding (concern that tamoxifen or acolbifene may be in breast milk) or nursing within the past 12 months (concern about milk fistula with RPFNA)
* Prior invasive breast cancer within the past 5 years
* Other prior invasive cancer > T1 stage (other than non-melanoma skin) within the past 5 years
* Pathogenic or likely pathogenic germline mutation in BRCA1/2 or PALB2 (These latter individuals are likely to undergo yearly ovarian screening and enlarging cysts could raise concern about ovarian cancer and lead to unnecessary diagnostic procedures)
* Type I or Type II diabetes mellitus requiring treatment with prescription medication
* Prior deep vein thrombosis, pulmonary embolus, or stroke
* History of chronic liver disease including NASH (nonalcoholic steatohepatitis) and chronic hepatitis C
* History of chronic hepatitis B or hepatitis C (danger of exacerbation of liver damage from hepatitis or tamoxifen-induced non-alcoholic fatty liver disease or non-alcoholic steatohepatitis)
* History of human immunodeficiency virus (HIV)-infection (danger of exacerbation of underlying clinically inapparent liver damage caused by HIV and/or hepatotoxicity can be induced by interaction of tamoxifen-induced CYP3A4 with direct anti-hepatitis C virus [HCV] agents)
* Current use of prescription anticoagulants such as Coumadin (warfarin), direct-acting oral anticoagulants such as Xarelto (rivaroxaban) or Eliquis (apixaban), or heparin
* Women who would not be able to or do not wish to discontinue daily use of aspirin (81 mg or higher) and aspirin containing products (81 mg or higher) at least 3 weeks prior to each RPFNA are not eligible. Women who would be able to stop daily use of aspirin and aspirin containing products at least 3 weeks prior to each RPFNA are eligible

  * NOTE: Women may resume daily use of aspirin and aspirin containing products 3 days after each RPFNA procedure
* Starting or stopping oral contraceptives (OCs) or hormonal progestin IUDs within 8 weeks of baseline RPFNA
* Current use or use within the prior 8 weeks of progesterone/progestin injections or progestin implants (due to concerns about high levels of progestin and lack of safety and efficacy data with low dose tamoxifen)
* Current use of other investigational agents
* Prior treatment with acolbifene for more than 2 months
* Prior treatment with tamoxifen for more than 2 months
* Current use of prescription immunosuppressive drugs
* History of allergic reactions attributed to tamoxifen or acolbifene or compounds of similar chemical composition
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2027-08-23 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in the relative abundance of the specific sequence of messenger ribonucleic acid that codes for AGR2 | Baseline up to 6 months
  Will be assessed in benign breast tissue acquired by random periareolar fine-needle aspiration. Change over the intervention period is expressed as the ratio of the relative abundance values (6-month value: baseline value) and then this fold change value is log transformed (base 2) for analysis. For this variable, values of zero indicate no change in the relative abundance of AGR2; positive values indicate an increase in the relative abundance; and negative values a decrease in the relative abundance.

SECONDARY OUTCOMES:
Change in Estrogen Response Gene Index (ERGI) | Baseline up to 6 months
  The genes assayed for this index are: ESR1, ESR2, GREB1, progesterone receptor (PGR), and TFF1. The log2-transformed values of the ratio of relative abundance (6-month value: baseline value) for GREB1, PGR, TFF1, and the ratio of ESR1:ESR2 are averaged to produce the ERGI. In cases where a specific gene or ratio cannot be evaluated for change over time, it is omitted from the average.
Relative change in mammographic absolute fibroglandular volume | Baseline up to 6 months
  Will be assessed via the completely automated Volpara™ software program. This will be performed from Digital Imaging and Communications in Medicine image files analyzed on a Research Server to which the Volpara™ algorithm has been loaded. The Volpara™ score card with volumetric assessments will be automatically generated. The volumetric measures may be less susceptible to technical variance (such as compression) than area of density.
Relative change in mammographic percentage (%) dense volume | Baseline up to 6 months
  Will be assessed via the completely automated Volpara™ software program. This will be performed from Digital Imaging and Communications in Medicine image files analyzed on a Research Server to which the Volpara™ algorithm has been loaded. The Volpara™ score card with volumetric assessments will be automatically generated. The volumetric measures may be less susceptible to technical variance (such as compression) than area of density.
Change in Menopause-Specific Quality of Life (MENQOL) | Baseline up to 6 months
  The responses to the 32 questions (will ask about symptoms over prior week) are clustered into four domains (vasomotor, psychosocial, physical, sexual). Worsening of problems (higher scores) over the course of the intervention will assessed by average scores for each of the four individual domains as well as the total MENQOL score.
Change in Hot Flash Score | Baseline up to 6 months
  The Hot Flash Score uses the product of the average number of hot flash/night sweat episodes per day and the average intensity (0= N/A, not experienced; 1= Mild; 2= Moderate; 3= Severe; 4= Very Severe).

CONTACTS AND LOCATIONS:
Overall Officials: Carol J Fabian, Principal Investigator — University of Kansas Medical Center
Locations (4):
- United States (4):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Northwestern University, Chicago, Illinois
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm